CLINICAL TRIAL: NCT06083363
Title: Longitudinal Recovery Trajectories After an Acute Respiratory Distress Syndrome, a New Understanding. The TENACITY Study
Brief Title: Longitudinal Recovery Trajectories After an Acute Respiratory Distress Syndrome, a New Understanding
Acronym: TENACITY
Status: Recruiting | Type: Observational
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Jessica González Gutiérrez MD, PhD, Medical Doctor, Doctor of Philosophy, Institut de Recerca Biomèdica de Lleida
Other Study IDs: PI23/01381
Record Dates: First submitted 2023-09-04; First posted 2023-10-16 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: ARDS; ARDS Disease Progression
Keywords: ARDS; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Per visit:
  2 EDTA Tubes (6ml)
  1 Tempus RNS tube (2,5ml)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-ICU with ARDS: Patients admitted to the ICU who have developed Acute Respiratory Distress Syndrome (ARDS), as defined according the new 2023 guidelines (Matthay et.al, 2023)
- post-ICU without ARDS: Patients admitted to the ICU who have suffered a severe pneumonia, needing advanced respiratory support, but without developing ARDS according to the new 2023 guidelines.

SUMMARY:
COVID-19 resulted in the largest cohort of critical illness survivors in history, heightened awareness of the importance of the respiratory sequelae after an acute distress respiratory syndrome (ADRS). Despite the advancement of acute-phase ARDS management, it is unknown whether there are differences in the longitudinal recovery trajectories between patients with post-ARDS due to COVID-19 and due to other causes. The main objective of the study is to identify risk factors of pulmonary sequela (lung diffusing capacity) at long-term follow-up in survivors of ARDS. The investigators are also interested in describing the long-term longitudinal recovery trajectories at a multi-dimensional level (symptoms, quality of life, neurocognitive, other lung function parameters, exercise capacity, chest imaging and molecular profiles) of ARDS survivors, and compared between ARDS caused by COVID-19. The ultimate goal is to understand the pathobiological mechanisms associated with a severe lung injury at the long term, allowing the introduction of clinical guidelines for the management of post-ARDS patients and the assignment of personalized interventions.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) resulted in the largest cohort of critical illness survivors in history, heightened awareness of the importance of the multi-dimensional sequelae after an acute distress respiratory syndrome (ADRS). With the advancement of acute-phase ARDS management, it is unknown whether there are differences in longitudinal recovery trajectories in terms of lung function, symptoms, quality of life, neurocognitive disorders, exercise capacity, chest imaging, and even at molecular basis between patients with post-ARDS due to COVID-19 and due to other causes. This project will continue to generate information about non-COVID-19 post-ARDS based on the experience in our post-COVID consultation that began in May 2020.

The main objective of the study is to identify risk factors of pulmonary sequela in terms of DLCO at long-term follow-up in survivors of ARDS. The investigators are also interested in describing the long-term longitudinal recovery trajectories at a multidimensional level (symptoms, quality of life, neurocognitive, other lung function parameters, exercise capacity, chest imaging and molecular profiles) of ARDS survivors. Furthermore, risk factors as well as recovery trajectories will be compared between ARDS caused by COVID-19 and non-COVID-19. The ultimate goal is to understand the pathobiological mechanisms associated with a severe lung injury at the long term (one year after hospital discharge), in order to provide novel therapeutic targets to develop future intervention studies.

For doing so, adult ARDS survivors of any origin (different than COVID-19) (n=246) referred to the post-CRITICAL consultation at the University Hospitals of Arnau de Vilanova and Santa Maria (Lleida), University Hospital Joan XXIII (Tarragona) and Verge de la Cinta (Tortosa) will be included in this multicentric, prospective, longitudinal and observational study. Previous standardized protocol will be followed at 3, 6 and 12 months after hospital discharge with a complete evaluation of symptoms, neurocognitive, memory problems and quality of life. Lung function, exercise test, chest CT and molecular analysis will be performed at each time point. The prognostic factors and the longitudinal recovery trajectories of ARDS survivors will be assessed using latent class mixed and machine learning artificial models.

The specific objectives to achieve the general objective are the following:

* Objective 1: To identify risk factors of lung function sequelae (spirometry, total lung volumes and lung diffusing capacity) in non-COVID-19 ARDS survivors.
* Objective 2: To identify risk factors of structural pulmonary sequelae (chest CT findings) in non-COVID-19 ARDS survivors.
* Objective 3: To identify risk factors of symptoms, neurocognitive disorders (BC-CCI, MOCA) and quality of life (SF-12) in non-COVID-19 ARDS survivors.
* Objective 4: To develop a clinical scoring tool to predict pulmonary sequelae at short- and long-term follow-up.
* Objective 5: To compare risk factors and recovery trajectories with COVID-19 ARDS survivors using data previously collected.
* Objective 6: To use artificial intelligence to identify multidimensional phenotypes associated with recovery trajectories.
* Objective 7: To design a cost-effective follow-up plan after hospital discharge in ARDS patients based on hospital risk factors.
* Objective 8: To identify molecular profiles according to recovery trajectories in non-COVID-19 ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥18 years
* Admission to the ICU
* Diagnosis of severe pneumonia and/or diagnosis of acute respiratory distress syndrome (ARDS) based on the 2023 definition due to any origin (infectious and non-infectious)

Exclusion Criteria:

* Life expectancy less than a year
* Transfer to another hospital during hospitalization or follow-up
* Stay in palliative care
* Severe mental disability that makes it impossible to carry out pulmonary function tests during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients admited to the intensive care unit of the 3 participant hospitals whot meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in lung diffusing capacity | 3, 6 and 12 months
  Changes in the results of lung diffusing capacity (DLCO) in terms of mL/mmHg/MI
Changes in lung diffusing capacity | 3, 6 and 12 months
  Changes in the results of lung diffusing capacity (DLCO) in terms of percentage (%)
Changes in lung volumes | 3, 6 and 12 months
  Changes in the results of lung capacity or total lung capacity (TLC) in terms of Liters (L)
Changes in lung volumes | 3, 6 and 12 months
  Changes in the results of lung capacity or total lung capacity (TLC) in terms of percentage (%)
Changes in chest CT findings | 3, 6 and 12 months
  Identification of structural pulmonary sequelae in terms of chest CT findings

SECONDARY OUTCOMES:
Changes in the perceived cognitive difficulties | 3, 6 and 12 months
  Changes in the results of the British Columbia Cognitive Complaints Inventory (BC-CCI) test.
  The scale consists of 6 items assessing perceived problems with concentration, memory, expressing thoughts, word finding, slow thinking, and difficulty solving problems in the past 7 days. Scores on each item (ranging from 0, not at all, to 3, very much) are summed to yield a total score ranging from 0 to 18; higher scores indicate greater severity of cognitive complaints.
Changes in the cognitive function | 3, 6 and 12 months
  Changes in the results of Montreal Cognitive Assessment (MoCA) test.
  The MoCA test examines seven domains of cognitive function with a total of 11 different exercises and tasks. The total score ranges from 0 to 30, lower scores indicate greater severity of cognitive impairment.
Changes in the fatigue status | 3, 6 and 12 months
  Changes in the results of Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4)
  This scale is a short test of 13-item that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is 0-52, being the higher the score, the better the quality of life and less perception of fatigue.
Changes in the levels of anxiety | 3, 6 and 12 months
  Changes in the results of Hospital Anxiety and Depression Scale (HAD)
  The scale determines the levels of anxiety and depression that a person is experiencing. It is a 14 item scale (7 of the items relate to anxiety and 7 relate to depression). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Lower scores indicate less anxiety or depression.
Changes in independence to carry out daily activities | 3, 6 and 12 months
  Changes in the results of Barthel test.
  Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living. The Index yields a total score out of 100 - the higher the score, the greater the degree of functional independence. This score is calculated by simply totaling the individual item scores.
Changes in the perception of life quality | 3, 6 and 12 months
  Changes in the results of 12-Item Short Form Survey (SF-12) test.
  The SF-12 is a self-reported outcome measure composed by 12 items which examine eight dimensions of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Validation of a clinical scoring tool | 3, 6 and 12 months
  Validation of a clinical scoring tool to predict pulmonary sequelae at short- and long-term follow-up.
Cost-effectiveness of a follow-up plan | 3, 6 and 12 months
  Only direct costs will be considered. Analysis will include an estimation of quality-adjusted life-years (QALYs) gained
Identification of molecular profiles | 3, 6 and 12 months
  Classification of the population in different molecular profiles according to their recovery trajectories
Multidimensional phenotypes | 3, 6 and 12 months
  multidimensional phenotypes associated with recovery trajectories defined with artificial intelligence
Recovery trajectories of lung diffusing capacity | 3, 6 and 12 months
  Comparison of risk factors and recovery trajectories in terms of lung diffusing capacity (DLCO) with COVID-19 ARDS survivors using data previously collected.
Recovery trajectories of total lung capacity | 3, 6 and 12 months
  Comparison of risk factors and recovery trajectories in terms of total lung capacity (TLC) with COVID-19 ARDS survivors using data previously collected.
Recovery trajectories of perception of life quality | 3, 6 and 12 months
  Comparison of risk factors and recovery trajectories in terms of perception of life quality (SF12 test) with COVID-19 ARDS survivors using data previously collected.
Recovery trajectories of perception of fatigue | 3, 6 and 12 months
  Comparison of risk factors and recovery trajectories in terms of perception of fatigue (FACIT-4 test) with COVID-19 ARDS survivors using data previously collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica González Gutiérrez, MD, PhD, Principal Investigator — Institut de Recerca Biomèdica de Lleida
Locations (3):
- Spain (3):
  - Hospital de Tortosa Verge de la Cinta, Tortosa, Tarragona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitari Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No